CLINICAL TRIAL: NCT01171183
Title: Clinical Efficacy of Carvedilol for Psychostimulant Dependence
Brief Title: Carvedilol for Psychostimulant Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2P50DA018197 (NIH); 2P50DA018197 (NIH)
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Cocaine Dependence; Cocaine Withdrawal
Keywords: cocaine dependence; cocaine withdrawal
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Carvedilol controlled release (Active Comparator): controlled release carvedilol (Coreg CR) at 80 mg/day in once daily dosing
  Interventions: Drug: controlled release carvedilol

INTERVENTIONS:
Drug: controlled release carvedilol — carvedilol (Coreg CR) 80 mg/day in once daily dosing for 12 weeks followed by a 2-week taper
  Other Names: Coreg CR
  Arms: Carvedilol controlled release
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study examines whether carvedilol prolongs abstinence in recently abstinent cocaine dependent participants.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Cocaine dependence, as assessed by the substance abuse section of the Structured Clinical Interview for DSM-IV.
* At least weekly self-reported cocaine use during a preceding three month period
* Urine toxicology screen positive for cocaine or cocaine metabolite
* Women of childbearing age must have a negative pregnancy test, agree to adequate contraception to prevent pregnancy during the study, agree to monthly pregnancy testing and not be nursing

Exclusion Criteria:

* Suicide attempts within the past 12 months or suicidal ideations or psychotic symptoms in the past 6 months as determined by a study physician.
* Current opioid, alcohol or sedative physical dependence or amphetamine dependence.
* Major cardiovascular disorder that contraindicates study participation (e.g., history of myocardial infarction, stroke, congestive heart failure, cardiac arrhythmia, significant hypertension [i.e., >170 SBP or >110 DBP] or an unstable medical condition (e.g., untreated bacterial infection) as determined by the study physician.
* Asthma or chronic obstructive pulmonary disease.
* History of schizophrenia, or bipolar type I disorder.
* Use of medications that would be expected to have major interaction with carvedilol (e.g., rifampin, cimetidine, digoxin, diuretics).
* Medical contraindication to receiving carvedilol (e.g., diabetes, severe bradycardia, bronchial asthma or other bronchospastic condition, 2nd or 3rd degree AV block, sick sinus rhythm, severe hepatic impairment, documented hypersensitivity to carvedilol).
* Patients currently taking selective serotonin re-uptake inhibitors, antipsychotics and antidepressants (e.g., amitriptyline and imipramine).
* Liver function tests (i.e., liver enzymes) greater than three times normal levels.
* Systolic blood pressure > 170 mmHg or < 90 mmHg, diastolic blood pressure > 110 mmHg or < 60 mmHg, or heart rate of > 110 beats/min or < 55 beats/min. Supine blood pressure of 100/65 mm Hg or lower, a seated blood pressure of 90/60 mm Hg or lower, or an orthostatic change of >20mm Hg systolic or 10 mm Hg diastolic on standing.
* Participants with estimated glomerular filtration rate < 30 ml/min.
* Pregnant or nursing female.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Residential Facility (Weeks 1-2)
Arm/Group | Placebo | Carvedilol Controlled Release
Started | 15 (Those who were admitted to the residential facility and received at least one dose of study med.) | 16 (Subjects receiving at least one dose of study med. One did not due to BP outside study parameters.)
Completed | 13 | 10
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — BP outside of study parameters | 0 | 3
Period: Outpatient Participation (Weeks 3-10)
Arm/Group | Placebo | Carvedilol Controlled Release
Started | 12 (One subject completed the residential stay but withdrew prior to starting the outpatient phase.) | 9 (One subject completed the residential stay but was discharged due to protocol noncompliance.)
Completed | 2 | 4
Not Completed | 10 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 7 | 3
Not completed — Use of contraindicated med: PI term | 1 | 0

BASELINE CHARACTERISTICS:
Population: Those who were admitted to the residential unit and received at least one dose of medication. The data for one person in the carvedilol arm was excluded from analyses as the person did not meet inclusion criteria for the study and was discharged by the third day.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Carvedilol Controlled Release | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 14 | 9 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 12 | 26
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Urine Toxicology Screens
Description: Treatment Effectiveness Score, defined by the # of cocaine negative urines during the outpatient phase of the study divided by the total number of urine samples (30) and then multiplied by 100.
Time Frame: based on thrice weekly urine results during the 10-week outpatient phase
Population: Those who completed the residential facility and attended at least one outpatient clinic visit to complete assessments.
Measure: Mean (Standard Deviation); unit: percentage of cocaine negative urines
Arm/Group | Placebo | Carvedilol Controlled Release
Number analyzed (Participants) | 12 | 9
percentage of cocaine negative urines | 38.33 (35.23) | 41.85 (40.73)
Statistical Analysis 1: Comparison: Placebo vs Carvedilol Controlled Release; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; Median Difference (Final Values) = 3.52, Standard Deviation 37.64

2. Secondary Outcome: Retention
Description: number of weeks each participant is on study protocol
Time Frame: 12 weeks
Population: Those eligible participants who entered the residential facility and received at least one dose of study medication. One person in the carvedilol group is excluded from all analyses due to not meeting inclusion criteria.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Placebo | Carvedilol Controlled Release
Number analyzed (Participants) | 15 | 15
Weeks | 5.70 (4.04) | 5.28 (5.00)
Statistical Analysis 1: Comparison: Placebo vs Carvedilol Controlled Release; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.73, Standard Deviation 4.54

ADVERSE EVENTS:
Time Frame: during the 12 week trial as well as during the taper period
Arm/Group | Placebo | Carvedilol Controlled Release
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 8/15 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Carvedilol Controlled Release (N=15)
Severe disabling hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Severe disabling hip pain that was later found to be cancer that that metastasized to the hip
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Carvedilol Controlled Release (N=15)
lightheaded/dizzy (Vascular disorders) | 0 (0) | 3 (4)
dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
sleep disturbances (Nervous system disorders) | 1 (1) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
vaginal yeast infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
cold hand, tingling fingers (Nervous system disorders) | 1 (1) | 0 (0)
Penile discharge, burning (Renal and urinary disorders) | 1 (1) | 0 (0)
Night Sweats (Renal and urinary disorders) | 0 (0) | 1 (1)
cold symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — e.g., sore throat, swollen glands and congestion
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
nausea/vomiting and/or diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
flu-like symptoms (Immune system disorders) | 0 (0) | 1 (1) — e.g., body aches, vomiting, low energy
burned hand (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
swollen eye (Eye disorders) | 0 (0) | 1 (1)
numbness in hand (Nervous system disorders) | 1 (1) | 0 (0)
tiredness, lethargic (General disorders) | 1 (1) | 1 (1)
Anxious, restless (Psychiatric disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fell down (General disorders) | 0 (0) | 1 (1)
Sharp pain upper left torso (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Feeling "high" (Psychiatric disorders) | 1 (1) | 0 (0)
Paranoid delusions (Psychiatric disorders) | 1 (1) | 0 (0)
Frequent urination (Renal and urinary disorders) | 1 (1) | 0 (0)
Insect bite (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Elevated blood pressure (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small numbers of participants analyzed. Primary outcome measure based on successfully transition to outpatient phase of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No